CLINICAL TRIAL: NCT06954376
Title: Hyperbaric Oxygen Therapy as a Neuroprotective Intervention in Pediatric Acquired Brain Injury With Cognitive Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Abdel Hamid Gaml, Assistant Lecturer of Pediatrics, Faculty of Medicine, Kafr Elsheikh University, Kafr Elsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-137.
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hyperbaric Oxygen Therapy; Neuroprotective; Pediatric; Acquired Brain Injury; Cognitive Disability
MeSH Terms: conditions — Brain Injuries | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygen therapy group (Experimental): Patients received hyperbaric oxygen therapy (HBOT) using a monochamber hyperbaric chamber in addition to conventional rehabilitation.
  Interventions: Other: Hyperbaric oxygen therapy
- Control group (Active Comparator): Patients received conventional rehabilitation alone.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Hyperbaric oxygen therapy — Patients received hyperbaric oxygen therapy (HBOT) using a monochamber hyperbaric chamber in addition to conventional rehabilitation.
  Arms: Hyperbaric oxygen therapy group
Other: Conventional rehabilitation — Patients received conventional rehabilitation alone.
  Arms: Control group

SUMMARY:
This research aimed to investigate the effectiveness of hyperbaric oxygen therapy as a neuroprotective strategy for improving neurological outcomes in pediatric patients who have sustained acquired brain injury.

DETAILED DESCRIPTION:
Hyperbaric oxygen therapy (HBOT) is a medical treatment that delivers high-concentration oxygen in a pressurized chamber. It was developed initially from diving physiology research and popularized by Dutch surgeon Boerema for its life-sustaining plasma oxygen diffusion under hyperbaric conditions.

The fundamental mechanism of HBOT operates through Henry's Law, enabling unprecedented increases in tissue oxygen partial pressures that surpass levels achievable in normal atmospheric conditions.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 4-12 years with acquired brain injury.
* Confirmed neurological sequelae (e.g., cardiac arrest, intracranial hemorrhage, central nervous system infections, stroke, tumor, hypoxia) via MRI/neurological exam.

Exclusion Criteria:

* Positive family history of degenerative brain insults.
* Behavioral problems.
* Hyperbaric oxygen therapy contraindications:

  * Active epilepsy.
  * Respiratory insufficiency.
  * Uncontrolled heart failure.
  * Eustachian tube dysfunction.
  * Tympanic membrane rupture.
  * Mechanical ventilation dependency.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Communication Function Classification System | Eight months post-intervention
  The Communication Function Classification System (CFCS) was implemented to assess cognitive and speech capabilities across five levels of communicative competence.
  * Level I: Effective bidirectional communication (no need for external aids).
  * Level II: Consistent communication with familiar partners, occasional need for aids.
  * Level III: Communication requires significant effort and aids with familiar partners.
  * Level IV: Minimal communication, even with familiar partners.
  * Level V: No effective communication.

SECONDARY OUTCOMES:
Nutritional intake functionality | Eight months post-intervention
  Nutritional intake functionality was evaluated utilizing the Functional Oral Intake Scale (FOIS). This seven-point scale was structured to differentiate between tube-dependent nutrition and total oral intake capabilities.
  * Level 1: Tube-dependent, no oral intake.
  * Level 2: Tube-dependent, minimal oral intake (e.g., ice chips).
  * Level 3: Tube-dependent, inconsistent oral intake of pureed foods.
  * Level 4: Oral intake of pureed foods only.
  * Level 5: Oral intake of soft foods.
  * Level 6: Oral intake of regular diet with modifications.
  * Level 7: Unrestricted oral intake (regular diet).
Visual function assessment | Eight months post-intervention
  Visual function assessment was conducted through visual evoked potential testing, providing objective measurements of visual pathway integrity. Neurodevelopmental status was comprehensively evaluated using the Griffiths Mental Development Scales (GMDS). The GMDS yielded both subscale scores and an overall General Quotient (GQ).
  * ≥90: Normal development.
  * 80-89: Mild disability.
  * 70-79: Moderate disability.
  * <70: Severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.